CLINICAL TRIAL: NCT01891344
Title: A Phase 2, Open-Label Study of Rucaparib in Patients With Platinum-Sensitive, Relapsed, High-Grade Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer (ARIEL2)
Brief Title: A Study of Rucaparib in Patients With Platinum-Sensitive, Relapsed, High-Grade Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer (ARIEL2)
Acronym: ARIEL2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Collaborators: Foundation Medicine (Industry); Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-017; 2013-000517-20 (EudraCT Number)
Record Dates: First submitted 2013-06-20; First posted 2013-07-03 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: ovarian cancer; fallopian tube cancer; primary peritoneal cancer; peritoneal cancer; platinum sensitive; relapsed disease; PARP Inhibitor; rucaparib; homologous recombination; homologous recombination deficiency; genomic scarring; loss of heterozygosity; CO-338; PF 01367338; AG 14699; platinum sensitive ovarian cancer; platinum sensitive fallopian tube cancer; platinum sensitive primary peritoneal cancer; platinum sensitive peritoneal cancer; gynecological cancer; Clovis; Clovis Oncology; ARIEL2; ARIEL 2; ARIEL3; ARIEL 3
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Recurrence | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ovarian cancer (Experimental): rucaparib
  Interventions: Drug: Oral rucaparib

INTERVENTIONS:
Drug: Oral rucaparib — 600 mg BID
  Other Names: CO-338; PF 01367338; AG 14699

SUMMARY:
The purpose of this study is to determine which patients with ovarian, fallopian tube, and primary peritoneal cancer will best respond to treatment with rucaparib.

DETAILED DESCRIPTION:
Rucaparib is an orally available, small molecule inhibitor of poly-adenosine diphosphate [ADP] ribose polymerase (PARP) being developed for treatment of ovarian cancer associated with homologous recombination (HR) DNA repair deficiency (HRD). The safety and efficacy of rucaparib has been evaluated in several Phase 1 and Phase 2 studies. An oral formulation is the focus of current development efforts. Rucaparib is currently being investigated as monotherapy in patients with cancer associated with breast cancer susceptibility gene 1 (BRCA1) or BRCA2 mutations.

Clinical data with PARP inhibitors indicate there is an ovarian cancer patient population beyond just those with germline BRCA (gBRCA) mutations that may benefit from treatment with a PARP inhibitor. This study will define a molecular signature of HRD in ovarian cancer that correlates with response to rucaparib and enables selection of appropriate ovarian cancer patients for treatment with rucaparib. The HRD signature will be based on an association between the extent of genomic scarring (a downstream consequence of HRD) in a patient's tumor and observed clinical benefit from rucaparib treatment. Genomic scarring can be assessed by quantifying the extent of loss of heterozygosity across the tumor genome (tumor genomic LOH). One of the main advantages of detecting tumor genomic LOH is that it can identify HRD tumors regardless of the underlying mechanisms, which include both known (i.e., BRCA mutations) and unknown genetic and other mechanisms.

Once determined, this signature will be prospectively applied to ARIEL2 PART 2 and ARIEL3. This Phase 2 study (ARIEL2) will also compare archival versus recently collected tumor tissue in order to validate the use of archival tumor tissue for assessment of HRD status in ARIEL3.

This study will include 2 parts:

PART 1 (completed enrollment): Evaluation of HRD status and rucaparib efficacy in patients who received ≥1 prior platinum-based regimen and had platinum-sensitive disease

PART 2 (completed enrollment): Evaluation of HRD status and rucaparib efficacy in patients who received at least 3 prior chemotherapy regimens

ELIGIBILITY:
The following eligibility criteria pertain to patients enrolling into PART 2 of the study:

Inclusion:

* Have a histologically confirmed diagnosis of high grade serous or Grade 2 or Grade 3 endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Received at least 3 prior chemotherapy regimens. Non-chemotherapy regimens and maintenance therapies administered as single agent treatment will not count as a chemotherapy regimen
* Relapsed/progressive disease as confirmed by CT scan
* Have biopsiable and measurable disease. Note: biopsy is optional for patients known to harbor a deleterious gBRCA mutation
* Have sufficient archival formalin-fixed paraffin-embedded (FFPE) tumor tissue available for planned analyses

Exclusion:

* History of prior cancers except for those that have been curatively treated, with no evidence of cancer currently (provided all chemotherapy was completed >6 months prior and/or bone marrow transplant >2 years prior to first dose of rucaparib).
* Prior treatment with any PARP inhibitor
* Symptomatic and/or untreated central nervous system metastases
* Pre-existing duodenal stent and/or any other gastrointestinal disorder or defect that would, in the opinion of the Investigator, interfere with absorption of rucaparib
* Hospitalization for bowel obstruction within 3 months prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- United States (36):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arizona Cancer Center, Tucson, Arizona
  - Saint Jude Heritage Medical Center, Fullerton, California
  - University of California Los Angeles, Los Angeles, California
  - UC San Diego, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Medical Oncology, Santa Maria, California
  - Stanford University, Stanford, California
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - University of Miami Hospital & Clinics Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - UF Health Cancer Center, Orlando, Florida
  - Horizon BioAdvance, Lafayette, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Women's Cancer Care Associates, Albany, New York
  - New York University Langone Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hope - A Woman's Cancer Institute, Asheville, North Carolina
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (8):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Flinders Cancer Clinic - Flinders Medical Centre (FMC), Bedford Park, South Australia
  - Mercy Hospital for Women, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Crown Princess Mary Cancer Centre (Westmead Hospital), Westmead, Wentworthville
  - Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (11):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Centre, Edmonton, Alberta
  - British Columbia Cancer Agency, Kelowna, British Columbia
  - BC Cancer Agency - Fraser Valley Centre, Surrey, British Columbia
  - Vancouver Cancer Centre, British Columbia Cancer Agency (BCCA), Vancouver, British Columbia
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec
- France (8):
  - Institut Bergonie, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Institut Claudius Regaud, Toulouse, Midi-Pyrenees
  - Centre Catherine de Sienne, Nantes, Pays de la Loire Region
  - Hopital Tenon, Paris, Île-de-France Region
  - Hôpital Européen Georges-Pompidou, Paris, Île-de-France Region
  - Institut de cancerologie Gustave Roussy, Villejuif, Île-de-France Region
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Instituto Valencia de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (9):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Royal Marsden Sutton Hospital, Sutton, Surrey
  - St James University Hospital, Leeds, West Yorkshire
  - Addenbrooke's Hospital, Cambridge
  - Royal Marsden NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London
  - University College London, London
  - The Christie NHS Foundation Trust, Manchester
  - Sir Bobby Robson Cancer Trials Research Centre, Northern Centre for Cancer Care, Newcastle upon Tyne

REFERENCES:
- [Derived] Green ML, Ma SC, Goble S, Giordano H, Maloney L, Simmons AD, Beltman J, Harding TC, Xiao JJ. Population pharmacokinetics of rucaparib in patients with advanced ovarian cancer or other solid tumors. Cancer Chemother Pharmacol. 2022 May;89(5):671-682. doi: 10.1007/s00280-022-04413-7. Epub 2022 Apr 10. PMID 35397664
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Swisher EM, Kwan TT, Oza AM, Tinker AV, Ray-Coquard I, Oaknin A, Coleman RL, Aghajanian C, Konecny GE, O'Malley DM, Leary A, Provencher D, Welch S, Chen LM, Wahner Hendrickson AE, Ma L, Ghatage P, Kristeleit RS, Dorigo O, Musafer A, Kaufmann SH, Elvin JA, Lin DI, Chambers SK, Dominy E, Vo LT, Goble S, Maloney L, Giordano H, Harding T, Dobrovic A, Scott CL, Lin KK, McNeish IA. Molecular and clinical determinants of response and resistance to rucaparib for recurrent ovarian cancer treatment in ARIEL2 (Parts 1 and 2). Nat Commun. 2021 May 3;12(1):2487. doi: 10.1038/s41467-021-22582-6. PMID 33941784
- [Derived] Kristeleit RS, Oaknin A, Ray-Coquard I, Leary A, Balmana J, Drew Y, Oza AM, Shapira-Frommer R, Domchek SM, Cameron T, Maloney L, Goble S, Lorusso D, Ledermann JA, McNeish IA. Antitumor activity of the poly(ADP-ribose) polymerase inhibitor rucaparib as monotherapy in patients with platinum-sensitive, relapsed, BRCA-mutated, high-grade ovarian cancer, and an update on safety. Int J Gynecol Cancer. 2019 Nov;29(9):1396-1404. doi: 10.1136/ijgc-2019-000623. PMID 31685558
- [Derived] Swisher EM, Lin KK, Oza AM, Scott CL, Giordano H, Sun J, Konecny GE, Coleman RL, Tinker AV, O'Malley DM, Kristeleit RS, Ma L, Bell-McGuinn KM, Brenton JD, Cragun JM, Oaknin A, Ray-Coquard I, Harrell MI, Mann E, Kaufmann SH, Floquet A, Leary A, Harding TC, Goble S, Maloney L, Isaacson J, Allen AR, Rolfe L, Yelensky R, Raponi M, McNeish IA. Rucaparib in relapsed, platinum-sensitive high-grade ovarian carcinoma (ARIEL2 Part 1): an international, multicentre, open-label, phase 2 trial. Lancet Oncol. 2017 Jan;18(1):75-87. doi: 10.1016/S1470-2045(16)30559-9. Epub 2016 Nov 29. PMID 27908594
- See also: ARIEL trials website — http://arielstudy.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 491 subjects were recruited from 64 sites across 6 countries.
Groups:
- Part 1: tBRCA: Patients with a deleterious BRCA (breast cancer susceptibility gene) mutation detected in their tumor. Part 1 enrolled patients who received ≥ 1 prior platinum-based regimen and had platinum-sensitive disease.
- Part 1: Non-tBRCA LOH+: Patients without a BRCA mutation in their tumor, but have high LOH (loss of heterozygosity). Part 1 enrolled patients received ≥ 1 prior platinum-based regimen and had platinum-sensitive disease.
- Part 1: Non-tBRCA LOH-: Patients without a BRCA mutation in their tumor, but have low LOH. Part 1 enrolled patients received ≥ 1 prior platinum-based regimen and had platinum-sensitive disease.
- Part 1: Non-tBRCA LOH Unknown: Patients without a BRCA mutation in their tumor, and have unknown LOH due to missing results and/or failed test result(s). Part 1 enrolled patients received ≥ 1 prior platinum-based regimen and had platinum-sensitive disease.
- Part 2: tBRCA: Patients with a deleterious BRCA mutation detected in their tumor. Part 2 enrolled patients who received at least 3, but no more than 4, prior chemotherapy regimens.
- Part 2: Non-tBRCA LOH+: Patients without a BRCA mutation in their tumor, but have high LOH. Part 2 enrolled patients who received at least 3, but no more than 4, prior chemotherapy regimens.
- Part 2: Non-tBRCA LOH-: Patients without a BRCA mutation in their tumor, but have low LOH. Part 2 enrolled patients who received at least 3, but no more than 4, prior chemotherapy regimens.
- Part 2: Non-tBRCA LOH Unknown: Patients without a BRCA mutation in their tumor, and have unknown LOH due to missing results and/or failed test result(s). Part 2 enrolled patients who received at least 3, but no more than 4, prior chemotherapy regimens.
Period: Overall Study
Arm/Group | Part 1: tBRCA | Part 1: Non-tBRCA LOH+ | Part 1: Non-tBRCA LOH- | Part 1: Non-tBRCA LOH Unknown | Part 2: tBRCA | Part 2: Non-tBRCA LOH+ | Part 2: Non-tBRCA LOH- | Part 2: Non-tBRCA LOH Unknown
Started | 40 | 82 | 70 | 12 | 84 | 73 | 107 | 23
Completed | 34 | 80 | 70 | 11 | 80 | 72 | 107 | 23
Not Completed | 6 | 2 | 0 | 1 | 4 | 1 | 0 | 0
Not completed — Ongoing | 6 | 2 | 0 | 1 | 4 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- tBRCA: Patients with a deleterious BRCA mutation detected in their tumor.
- Non-tBRCA LOH+: Patients without a BRCA mutation in their tumor, but have high LOH.
- Non-tBRCA LOH-: Patients without a BRCA mutation in their tumor, but have low LOH.
- Non-tBRCA LOH Unknown: Patients without a BRCA mutation in their tumor, and have unknown LOH due to missing results and/or failed test result(s).
- Total: Total of all reporting groups
Arm/Group | tBRCA | Non-tBRCA LOH+ | Non-tBRCA LOH- | Non-tBRCA LOH Unknown | Total
Number analyzed (Participants) | 124 | 155 | 177 | 35 | 491
Age, Continuous [Median (Full Range); unit: years] — Population: Overall participant count is separated into Part 1 and Part 2 patients.
  years
    Part 1: number analyzed (Participants) | 40 | 82 | 70 | 12 | 204
    Part 1 | 58.5 [33 to 78] | 65 [39 to 83] | 65 [31 to 86] | 69.5 [44 to 81] | 64.5 [31 to 86]
    Part 2: number analyzed (Participants) | 84 | 73 | 107 | 23 | 287
    Part 2 | 60.5 [41 to 82] | 61 [35 to 82] | 64 [42 to 91] | 62 [43 to 81] | 63 [35 to 91]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Overall participant count is separated into Part 1 and Part 2 patients.
  Participants
    Part 1: number analyzed (Participants) | 40 | 82 | 70 | 12 | 204
    Part 1: Female | 40 | 82 | 70 | 12 | 204
    Part 1: Male | 0 | 0 | 0 | 0 | 0
    Part 2: number analyzed (Participants) | 84 | 73 | 107 | 23 | 287
    Part 2: Female | 84 | 73 | 107 | 23 | 287
    Part 2: Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall participant count is separated into Part 1 and Part 2 patients.
  Participants
    Part 1: number analyzed (Participants) | 40 | 82 | 70 | 12 | 204
    Part 1: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
    Part 1: Asian | 3 | 4 | 5 | 1 | 13
    Part 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Part 1: Black or African American | 1 | 2 | 1 | 1 | 5
    Part 1: White | 33 | 67 | 56 | 10 | 166
    Part 1: More than one race | 0 | 0 | 0 | 0 | 0
    Part 1: Unknown or Not Reported | 2 | 9 | 8 | 0 | 19
    Part 2: number analyzed (Participants) | 84 | 73 | 107 | 23 | 287
    Part 2: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
    Part 2: Asian | 5 | 4 | 5 | 0 | 14
    Part 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
    Part 2: Black or African American | 0 | 1 | 0 | 0 | 1
    Part 2: White | 59 | 46 | 82 | 18 | 205
    Part 2: More than one race | 0 | 0 | 0 | 0 | 0
    Part 2: Unknown or Not Reported | 19 | 22 | 19 | 5 | 65
Number of Prior Chemotherapy Regimens [Count of Participants; unit: Participants] — Population: Overall participant count is separated into Part 1 and Part 2 patients.
  Participants
    Part 1: number analyzed (Participants) | 40 | 82 | 70 | 12 | 204
    Part 1: 0 | 0 | 0 | 0 | 0 | 0
    Part 1: 1 | 17 | 45 | 47 | 10 | 119
    Part 1: 2 | 14 | 21 | 16 | 1 | 52
    Part 1: 3 | 4 | 13 | 6 | 1 | 24
    Part 1: 4 | 4 | 1 | 0 | 0 | 5
    Part 1: 5 | 1 | 1 | 1 | 0 | 3
    Part 1: >5 | 0 | 1 | 0 | 0 | 1
    Part 2: number analyzed (Participants) | 84 | 73 | 107 | 23 | 287
    Part 2: 0 | 0 | 0 | 0 | 0 | 0
    Part 2: 1 | 0 | 0 | 0 | 0 | 0
    Part 2: 2 | 0 | 1 | 1 | 0 | 2
    Part 2: 3 | 52 | 44 | 73 | 17 | 186
    Part 2: 4 | 32 | 28 | 31 | 6 | 97
    Part 2: 5 | 0 | 0 | 2 | 0 | 2
    Part 2: >5 | 0 | 0 | 0 | 0 | 0
Number of Prior Platinum Regimens [Count of Participants; unit: Participants] — Population: Overall participant count is separated into Part 1 and Part 2 patients.
  Participants
    Part 1: number analyzed (Participants) | 40 | 82 | 70 | 12 | 204
    Part 1: 0 | 0 | 0 | 0 | 0 | 0
    Part 1: 1 | 17 | 45 | 47 | 10 | 119
    Part 1: 2 | 15 | 25 | 16 | 1 | 57
    Part 1: 3 | 6 | 10 | 6 | 1 | 23
    Part 1: >3 | 2 | 2 | 1 | 0 | 5
    Part 2: number analyzed (Participants) | 84 | 73 | 107 | 23 | 287
    Part 2: 0 | 0 | 0 | 0 | 0 | 0
    Part 2: 1 | 2 | 4 | 7 | 3 | 16
    Part 2: 2 | 34 | 31 | 55 | 7 | 127
    Part 2: 3 | 40 | 36 | 44 | 12 | 132
    Part 2: >3 | 8 | 2 | 1 | 1 | 12
Platinum Sensitivity Status [Count of Participants; unit: Participants] — Refractory = Best response of progressive disease (PD) and PD occurs during or up to 2 months after regimen; Resistant = PD 0-<6 months after last platinum with best response other than PD; Sensitive = PD ≥6 months after last platinum Population: Overall participant count is separated into Part 1 and Part 2 patients.
  Participants
    Part 1: number analyzed (Participants) | 40 | 82 | 70 | 12 | 204
    Part 1: Refractory | 0 | 0 | 0 | 0 | 0
    Part 1: Resistant | 0 | 1 | 0 | 1 | 2
    Part 1: Sensitive | 40 | 81 | 70 | 11 | 202
    Part 2: number analyzed (Participants) | 84 | 73 | 107 | 23 | 287
    Part 2: Refractory | 12 | 14 | 18 | 4 | 48
    Part 2: Resistant | 41 | 46 | 56 | 15 | 158
    Part 2: Sensitive | 31 | 13 | 33 | 4 | 81

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) According to RECIST v1.1 in Molecularly-defined HRD (Homologous Recombination Deficiency) Subgroups (Part 1 of Study)
Description: The primary efficacy endpoint of PFS is calculated as 1+ the number of days from the first dose of study drug to disease progression by RECIST (Response Evaluation Criteria in Solid Tumors), as determined by the investigator or death due to any cause, whichever occurs first. Progression is defined using RECIST v1.1, as at least a 20% increase in the sum of the longest diameter of target lesions, or a measureable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Assessments every 8 weeks from C1D1 until disease progression, death or withdrawal of consent. After 18 months on study, assessments every 16 weeks. Total follow-up was up to approximately 3 years.
Population: Safety population by HRD subgroups: Consists of all Part 1 patients who received at least one dose of rucaparib.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Part 1: tBRCA: Patients with a deleterious BRCA mutation detected in their tumor.
- Part 1: Non-tBRCA LOH+: Patients without a BRCA mutation in their tumor, but have high LOH.
- Part 1: Non-tBRCA LOH-: Patients without a BRCA mutation in their tumor, but have low LOH.
- Part 1: Non-tBRCA LOH Unknown: Patients without a BRCA mutation in their tumor, and have unknown LOH due to missing results and/or failed test result(s).
Arm/Group | Part 1: tBRCA | Part 1: Non-tBRCA LOH+ | Part 1: Non-tBRCA LOH- | Part 1: Non-tBRCA LOH Unknown
Number analyzed (Participants) | 40 | 82 | 70 | 12
Days | 388 [273 to 448] | 174 [158 to 231] | 160 [110 to 188] | 223 [55 to 499]
Statistical Analysis 1: Comparison: Part 1: tBRCA vs Part 1: Non-tBRCA LOH-; Test type: Superiority; Cox Proportional Hazard = 0.273, 95% CI 2-sided [0.170 to 0.437]
Statistical Analysis 2: Comparison: Part 1: Non-tBRCA LOH+ vs Part 1: Non-tBRCA LOH-; Test type: Superiority; Cox Proportional Hazard = 0.610, 95% CI 2-sided [0.428 to 0.871]

2. Primary Outcome: Objective Response Rate (ORR) by RECIST v1.1 in Molecularly-defined HRD Subgroups (Part 2 of Study)
Description: The confirmed response rate by RECIST v1.1 is defined as the percentage of patients with a confirmed complete response (CR) or partial response (PR) on subsequent tumor assessment at least 28 days after first response documentation. Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: as for outcome 1
Population: Safety population by HRD subgroups: Consist of all Part 2 patients who received at least one dose of rucaparib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2: tBRCA: Patients with a deleterious BRCA mutation detected in their tumor.
- Part 2: Non-tBRCA LOH+: Patients without a BRCA mutation in their tumor, but have high LOH.
- Part 2: Non-tBRCA LOH-: Patients without a BRCA mutation in their tumor, but have low LOH.
- Part 2: Non-tBRCA LOH Unknown: Patients without a BRCA mutation in their tumor, and have unknown LOH due to missing results and/or failed test result(s).
Arm/Group | Part 2: tBRCA | Part 2: Non-tBRCA LOH+ | Part 2: Non-tBRCA LOH- | Part 2: Non-tBRCA LOH Unknown
Number analyzed (Participants) | 84 | 73 | 107 | 23
percentage of participants | 31.0 [21.3 to 42.0] | 6.8 [2.3 to 15.3] | 5.6 [2.1 to 11.8] | 13.0 [2.8 to 33.6]

3. Secondary Outcome: Objective Response Rate (ORR) by RECIST v1.1 (Part 1 of Study)
Description: The confirmed response rate by RECIST v1.1 is defined as the percentage of patients with a confirmed CR or PR on subsequent tumor assessment at least 28 days after first response documentation. Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: as for outcome 1
Population: Safety population by HRD subgroups: Consist of all Part 1 patients who received at least one dose of rucaparib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: tBRCA | Part 1: Non-tBRCA LOH+ | Part 1: Non-tBRCA LOH- | Part 1: Non-tBRCA LOH Unknown
Number analyzed (Participants) | 40 | 82 | 70 | 12
percentage of participants | 80.0 [64.4 to 90.9] | 28.0 [18.7 to 39.1] | 10.0 [4.1 to 19.5] | 33.3 [9.9 to 65.1]

4. Secondary Outcome: Objective Response Rate (ORR) by RECIST v1.1 and GCIG CA-125 Criteria
Description: The endpoint of ORR defined as the percentage of patients with a best response of CR or PR using RECIST v 1.1 or a response per Gynecologic Cancer InterGroup cancer antigen 125 (GCIG CA-125) criteria. Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. A response to CA-125 has occurred if there is at least a 50% decrease from baseline: 1. in a sample collected after initiation of study treatment AND 2. that is confirmed in a subsequent sample collected ≥21 days after the prior sample. The absolute value of this confirmatory sample must be ≤110% of the prior sample. The date when the first sample with a 50% decrease from baseline is observed is the date of the CA-125 response.
Time Frame: as for outcome 1
Population: Safety population by HRD subgroups: Consist of all Part 1 and Part 2 patients who received at least one dose of rucaparib.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part 1: tBRCA | Part 1: Non-tBRCA LOH+ | Part 1: Non-tBRCA LOH- | Part 1: Non-tBRCA LOH Unknown | Part 2: tBRCA | Part 2: Non-tBRCA LOH+ | Part 2: Non-tBRCA LOH- | Part 2: Non-tBRCA LOH Unknown
Number analyzed (Participants) | 40 | 82 | 70 | 12 | 84 | 73 | 107 | 23
percentage of patients | 87.5 [73.2 to 95.8] | 46.3 [35.3 to 57.7] | 21.4 [12.5 to 32.9] | 50.0 [21.1 to 78.9] | 54.8 [43.5 to 65.7] | 12.3 [5.8 to 22.1] | 13.1 [7.3 to 21.0] | 30.4 [13.2 to 52.9]

5. Secondary Outcome: Duration of Response Per RECIST v1.1
Description: Duration of response (DOR) for any confirmed RECIST CR or PR measured from the date of the first occurrence of a response until the first occurrence of progressive disease (PD) per RECIST. For patients who continued treatment post-progression, the first date of progression was used for the analysis. Any patients with an ongoing response were censored at the date of the last post-baseline scan. Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: as for outcome 1
Population: Efficacy population by HRD subgroups. The overall number of patients analyzed includes only patients with confirmed RECIST CR or PR.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: tBRCA | Part 1: Non-tBRCA LOH+ | Part 1: Non-tBRCA LOH- | Part 1: Non-tBRCA LOH Unknown | Part 2: tBRCA | Part 2: Non-tBRCA LOH+ | Part 2: Non-tBRCA LOH- | Part 2: Non-tBRCA LOH Unknown
Number analyzed (Participants) | 32 | 23 | 7 | 4 | 26 | 5 | 6 | 3
Days | 281 [194 to 393] | 329 [174 to 451] | 169 [141 to 260] | 225 [100 to 1454] | 176 [169 to 312] | 282 [111 to NA] — The upper limit of the confidence interval is not estimated due to insufficient number of participants with events. | 314 [169 to NA] — The upper limit of the confidence interval is not estimated due to insufficient number of participants with events. | 181 [169 to 224]

6. Secondary Outcome: Progression-free Survival (PFS) According to RECIST v1.1 in Molecularly-defined HRD Subgroups (Part 2 of Study)
Description: Progression-Free Survival (PFS) is calculated as 1+ the number of days from the first dose of study drug to disease progression by RECIST, as determined by the investigator or death due to any cause, whichever occurs first. Progression is defined using RECIST v1.1, as at least a 20% increase in the sum of the longest diameter of target lesions, or a measureable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 1
Population: Safety population by HRD subgroups: Consist of all Part 2 patients who received at least one dose of rucaparib.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 2: tBRCA | Part 2: Non-tBRCA LOH+ | Part 2: Non-tBRCA LOH- | Part 2: Non-tBRCA LOH Unknown
Number analyzed (Participants) | 84 | 73 | 107 | 23
Days | 223 [188 to 275] | 57 [54 to 112] | 113 [63 to 165] | 110 [56 to 154]

7. Secondary Outcome: Overall Survival (Part 2 of Study)
Description: Overall survival (OS) is defined as the number of days from the date of first dose of study drug to the date of death (due to any cause). Patients without a known date of death will be censored on the date the patient was last known to be alive.
Time Frame: All patients in Part 2 were followed for survival, subsequent therapy, and secondary malignancy every 12 weeks until death, loss to follow-up, withdrawal of consent from study or study closure, whichever happened first, up to 7 years.
Population: Safety population by HRD subgroups: Consist of all Part 2 patients who received at least one dose of rucaparib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: tBRCA | Part 2: Non-tBRCA LOH+ | Part 2: Non-tBRCA LOH- | Part 2: Non-tBRCA LOH Unknown
Number analyzed (Participants) | 84 | 73 | 107 | 23
Months | 22.7 [16.7 to 28.6] | 14.7 [10.8 to 19.8] | 13.3 [9.1 to 16.0] | 14.1 [7.4 to 20.1]

8. Secondary Outcome: Steady State Trough (Cmin) Level Rucaparib Concentrations
Description: Per protocol, the secondary PK endpoint, trough (Cmin) concentrations of rucaparib were summarized with descriptive statistics overall and by cycle in all patients with at least one PK sample collected. Blood samples for trough level PK analysis of rucaparib were drawn at the following timepoints only: on Day 15 of Cycle 1 and on Day 1 of Cycles 2, 3, and 4. Data for other timepoints is not available.
Time Frame: Cycle 1 Day 15 to Cycle 4 Day 1, or approximately 10 weeks
Population: All Part 1 and Part 2 patients with at least one PK sample collected
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 1 Overall: Includes all Part 1 patients
- Part 2 Overall: Includes all Part 2 patients
Arm/Group | Part 1 Overall | Part 2 Overall
Number analyzed (Participants) | 196 | 267
ng/mL
  Cycle 1 Day 15 | 2020.76 (1145.164) | 2276.37 (1587.586)
  Cycle 2 Day 1: number analyzed (Participants) | 186 | 242
  Cycle 2 Day 1 | 1652.27 (935.503) | 1689.83 (1039.953)
  Cycle 3 Day 1: number analyzed (Participants) | 159 | 174
  Cycle 3 Day 1 | 1557.32 (952.903) | 1552.09 (1054.346)
  Cycle 4 Day 1: number analyzed (Participants) | 142 | 149
  Cycle 4 Day 1 | 1530.41 (765.940) | 1629.14 (1026.999)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time informed consent was obtained until 28 days after last dose of study drug, approximately 5 years.
Description: If a subject experiences the same preferred term (system organ class) multiple times, then the subject will be counted only once for that preferred term (system organ class). Adverse Events were monitored/assessed without regard to the subgroups.
Groups:
- Part 1 Overall: All patients who participated in Part 1 who received at least one dose of rucaparib
- Part 2 Overall: All patients who participated in Part 2 who received at least one dose of rucaparib
Arm/Group | Part 1 Overall | Part 2 Overall
All-Cause Mortality (participants affected / at risk) | 2/204 | 18/287
Serious Adverse Events (participants affected / at risk) | 54/204 | 92/287
Other Adverse Events (participants affected / at risk) | 203/204 | 285/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Overall (N=204) | Part 2 Overall (N=287)
Anaemia (Blood and lymphatic system disorders) | 11 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 6
Granulocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Cardiac congestive failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Long QT syndrome congenital (Congenital, familial and genetic disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 6
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 7
Obstruction gastric (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 11 | 8
Subileus (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 9
Asthenia (General disorders) | 1 | 4
General physical health deterioration (General disorders) | 0 | 7
Hyperthermia (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 4
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic haematoma (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 4 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 4
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 5
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 10
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 3
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Overall (N=204) | Part 2 Overall (N=287)
Anaemia (Blood and lymphatic system disorders) | 72 | 122
Neutropenia (Blood and lymphatic system disorders) | 12 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 44
Abdominal distension (Gastrointestinal disorders) | 41 | 31
Abdominal pain (Gastrointestinal disorders) | 63 | 89
Abdominal pain lower (Gastrointestinal disorders) | 12 | 12
Abdominal pain upper (Gastrointestinal disorders) | 31 | 35
Ascites (Gastrointestinal disorders) | 12 | 12
Constipation (Gastrointestinal disorders) | 95 | 81
Diarrhoea (Gastrointestinal disorders) | 76 | 83
Dry mouth (Gastrointestinal disorders) | 11 | 12
Dyspepsia (Gastrointestinal disorders) | 24 | 20
Flatulence (Gastrointestinal disorders) | 13 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 15
Nausea (Gastrointestinal disorders) | 161 | 219
Stomatitis (Gastrointestinal disorders) | 25 | 15
Vomiting (Gastrointestinal disorders) | 92 | 125
Asthenia (General disorders) | 24 | 67
Chills (General disorders) | 16 | 8
Fatigue (General disorders) | 140 | 157
Influenza like illness (General disorders) | 11 | 6
Oedema peripheral (General disorders) | 21 | 38
Pyrexia (General disorders) | 29 | 31
Nasopharyngitis (Infections and infestations) | 15 | 13
Upper respiratory tract infection (Infections and infestations) | 27 | 10
Urinary tract infection (Infections and infestations) | 37 | 33
Alanine aminotransferase increased (Investigations) | 83 | 85
Aspartate aminotransferase increased (Investigations) | 74 | 92
Blood alkaline phosphatase increased (Investigations) | 19 | 24
Blood cholesterol increased (Investigations) | 14 | 13
Blood creatinine increased (Investigations) | 37 | 65
Neutrophil count decreased (Investigations) | 20 | 12
Platelet count decreased (Investigations) | 15 | 36
Weight decreased (Investigations) | 42 | 30
White blood cell count decreased (Investigations) | 13 | 12
Decreased appetite (Metabolism and nutrition disorders) | 85 | 110
Dehydration (Metabolism and nutrition disorders) | 16 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 19
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 | 29
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 24
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 21
Dizziness (Nervous system disorders) | 42 | 35
Dysgeusia (Nervous system disorders) | 88 | 93
Headache (Nervous system disorders) | 36 | 35
Lethargy (Nervous system disorders) | 13 | 5
Neuropathy peripheral (Nervous system disorders) | 11 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 2
Anxiety (Psychiatric disorders) | 14 | 17
Insomnia (Psychiatric disorders) | 23 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 68
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 6
Erythema (Skin and subcutaneous tissue disorders) | 7 | 16
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 30 | 18
Pruritis (Skin and subcutaneous tissue disorders) | 20 | 16
Rash (Skin and subcutaneous tissue disorders) | 21 | 13
Hot flush (Vascular disorders) | 15 | 10
Hypertension (Vascular disorders) | 18 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT01891344/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT01891344/SAP_001.pdf